CLINICAL TRIAL: NCT03399214
Title: A Phase Ib Study to Evaluate Safety and Efficacy Profiles of IOP Injection for Magnetic Resonance Imaging (MRI) Contrast Agent in Healthy Subjects.
Brief Title: Phase Ib, Administration the IOP Injection for MRI Contrast Agent in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IOP-CT-002
Record Dates: First submitted 2018-01-02; First posted 2018-01-16 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOP Injection, Phase 1b, Cohort 1 (Experimental): IV injection, 0.27 mg/kg
  Interventions: Drug: IOP Injection
- IOP Injection, Phase 1b, Cohort 2 (Experimental): IV injection, 0.54 mg/kg
  Interventions: Drug: IOP Injection

INTERVENTIONS:
Drug: IOP Injection — T1 and T2

SUMMARY:
The objective of the study is to assess the dose dependent changes in MRI signal intensity (SI) in liver after IOP Injection intravenous administration in healthy volunteers.

DETAILED DESCRIPTION:
Find the max. signal change after IOP administration

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥ 20 ~40 years, BMI=18~27.
2. The biochemistry test results, complete blood count (CBC) test results, urinalysis test results, coagulation time test results must within normal range or considered clinically normal by the clinical investigator at screening.
3. Male subjects must take reliable contraceptive method(s) during and after the study for a period of 14 days.
4. No screening of drug or alcohol abuse within one year prior to study enrollment.
5. Subjects are willing to comply with the protocol and sign informed consent form.

Exclusion Criteria:

1. Subjects have serious allergic history or known allergy to MRI contrast agent.
2. Subjects with HBV, HCV, HIV.
3. Imaging and/or functional abnormalities of liver and/or spleen.
4. Subjects have alcohol or caffeine consumption within 48 hours prior to the administration of study contrast agent.
5. Subjects have electronically, magnetically and mechanically activated implanted devices.
6. Subjects have participated in other investigational trials or receive any contrast agents within 28 days prior to study enrollment.
7. Subjects with active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal ulcers, or medical conditions that may significantly affect action, adequate absorption and elimination of investigational contrast agent.
8. Subjects have taken any food 6 hours prior to administration.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The Change of MRI SI (%) in vessels, liver, and spleen | Day1: within 60 mins after IOP administration
  The optimal imaging time of IOP injection for the maximum SI (%)

SECONDARY OUTCOMES:
The changes from baseline in hematology data | within 14 days
  Complete blood count and differential count, Reticulocyte count
The incidence of all treatment-related adverse events (TRAE) | within 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Rheun-Chuan Lee, MD, Principal Investigator — rclee@vghtpe.gov.tw
Locations (1):
- Taipei Veterans General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No